CLINICAL TRIAL: NCT04506489
Title: Access to Maternity and Risk Factors in a Non-consultant Population - Longitudinal and Prospective Exploratory Study (PROXIMA)
Brief Title: Access to Maternity and Risk Factors in a Non-consultant Population (PROXIMA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/434
Record Dates: First submitted 2020-07-20; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-04

CONDITIONS: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychological investigation
  Interventions: Other: Psychological investigation

INTERVENTIONS:
Other: Psychological investigation — Psychological tests, psychological interviews.

SUMMARY:
Characterize the psychic and medical disorders related to pregnancy and motherhood in a group of primiparous and primigratic women.

ELIGIBILITY:
Inclusion Criteria:

* primiparous and primigest women,
* Singleton pregnancy
* Consultant at the University Hospital of Besançon in gynecology / obstetrics department - initial consultation
* 25 to 45 years old,
* European culture and speaking French,
* Living in a relationship with the spouse
* Spontaneous pregnancy, without medical help
* Having agreed to the use of this medical data as part of this research and the completion of the self-questionnaires.
* Patients who benefit from a social security scheme

Exclusion Criteria:

* Termination of pregnancy or non-progressive pregnancy
* Prematurity of the child (Childbirth before 37 weeks)
* Maternal pathologies acquired during pregnancy
* Fetal diseases acquired during pregnancy
* Pregnancy of twins or triplets
* Any type of medical difficulties occurring during pregnancy (gestational diabetes, high blood pressure, threat of preterm delivery, preeclampsia, ...)
* Any type of difficulty occurring during childbirth for example, hemorrhage of maternal deliverance
* Birth by cesarean section Birth necessitating the use of instruments that led to the transfer of the baby to the neonatology unit or to the kangaroo unit
* At birth, baby's Apgar less than 7.
* Fetal death
* Childbirth that did not occur at the CHU maternity ward

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primiparous women without mental and obstetric disorders monitoring in the Besançon University Hospital, during their pregnancy and after their birth.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Self questionnaire : health, Anxiety, Postnatal, Body Satisfaction, , Bartholomew, RelationShip, Social , Perinatal, Family Relationship , parental stress, dyadic alliance, Parental Bonding , Prenatal attachment , birth experience | 3 to 4 months of pregnancy
  units (scale)
Self questionnaire : health, Anxiety, Postnatal, Body Satisfaction, , Bartholomew, RelationShip, Social , Perinatal, Family Relationship , parental stress, dyadic alliance, Parental Bonding , Prenatal attachment , birth experience | 8-9 months of pregnancy
  units (scale)
Self questionnaire : health, Anxiety, Postnatal, Body Satisfaction, , Bartholomew, RelationShip, Social , Perinatal, Family Relationship , parental stress, dyadic alliance, Parental Bonding , Prenatal attachment , birth experience | 15 days to 1 month after birth
  units (scale)
Self questionnaire : health, Anxiety, Postnatal, Body Satisfaction, , Bartholomew, RelationShip, Social , Perinatal, Family Relationship , parental stress, dyadic alliance, Parental Bonding , Prenatal attachment , birth experience | 3 months after birth
  units (scale)
Self questionnaire : health, Anxiety, Postnatal, Body Satisfaction, , Bartholomew, RelationShip, Social , Perinatal, Family Relationship , parental stress, dyadic alliance, Parental Bonding , Prenatal attachment , birth experience | 6 months after birth
  units (scale)

CONTACTS AND LOCATIONS:
Overall Officials: Mottet Nicolas, Dr, Principal Investigator — CHU Besançon
Locations (1):
- Mathilde Pointurier, Besançon, Franche Comté, France